CLINICAL TRIAL: NCT01141556
Title: Effects of High-dose Intravenous Selenium (Selenase®) on the Systemic Inflammatory Response Syndrome and Related Organ Dysfunction
Brief Title: Effects of High-dose Intravenous Selenium (Selenase®) in Adult Patients Subjected to Elective All-cause Heart Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 236/09
Record Dates: First submitted 2010-06-08; First posted 2010-06-10 (Estimated); Last update posted 2012-10-25 (Estimated); Status verified 2012-10

CONDITIONS: Heart; Surgery, Heart, Functional Disturbance as Result; Self Efficacy
Keywords: selenium; clinical outcome; heart surgery

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo (NaCl) i.v. intraoperatively, followed by an daily bolus of Placebo (NaCl) i.v. until discharge from ICU (no longer than 13 days)
  Interventions: Drug: Selenase
- Selenase (Active Comparator): Selenase Bolus 4000 microgram i.v. intraoperatively, followed by an daily bolus of Selenase 1000 microgram i.v. until discharge from ICU (no longer than 13 days)
  Interventions: Drug: Selenase

INTERVENTIONS:
Drug: Selenase — After enrollment, patients will be prospectively randomized into two groups: a placebo group without selenium and a group receiving a loading dose of selenium 4000 μg intraoperatively,followed by a daily dosage of 1000 μg until leaving the ICU (longest supplementation 13 days).
  Other Names: Selenase: Selenium

SUMMARY:
Selenoenzymes play a major role in protecting cells against lipid peroxidation and they are involved in the inflammatory response regulation. The degree of selenium deficiency correlates with disease severity and the incidence of mortality in critically ill patients. The aim of our study is to evaluate, if high dosis selenium supplementation (loading dose 4000 μg, daily dosage 1000 μg) results in a significant reduction of inflammation-induced organ dysfunction and length of ICU-stay in patients after heart surgery.

DETAILED DESCRIPTION:
Selenium is a essential micronutrient that is present in form of selenocysteine in many enzymes. Selenoenzymes play a major role in protecting cells against lipid peroxidation and they are involved in the inflammatory response regulation. The degree of selenium deficiency correlates with disease severity and the incidence of mortality. Different studies showed that selenium supplementation had beneficial effects in critically ill patients with systemic inflammatory response syndrome (SIRS), reducing the rate of infectious complications and length of hospital stay.

Heart surgery is associated with a complex systemic inflammatory response and the extent correlates with the development of postoperative complications. Former clinical trials used selenium supplementation with a loading dose of normally 1000 to 2000 μg, followed by a daily dosage of 1000 μg. With these dosage regimes pharmacological investigations demonstrated a delayed increase of the selenium concentration in plasma and whole blood. As a result a delayed increase of selenoenzymes can be assumed.

Aim of our study is to evaluate, if high dosis selenium supplementation (loading dose 4000 μg, daily dosage 1000 μg) results in a significant reduction of inflammation-induced organ dysfunction and length of ICU-stay in patients after heart surgery.

Primary endpoints are: Clinical outcome quantified by using the Sequential Organ Failure Assessment (SOFA) Score and the length of ICU stay in hours.

Secondary endpoints are: incidence of acute renal failure, total requirement of vasoconstrictors and fluid replacement therapy

Inclusion criteria: written informed consent, males and females age ≥ 18 years, patients undergoing an elective heart surgery, normal renal function (serum creatinine ≤ 200 μmol/l)

Exclusion criteria: pregnancy, lack of written concent, emergency operation

ELIGIBILITY:
Inclusion Criteria:

* written informed consent
* males and females age ≥ 18 years
* patients undergoing an elective heart surgery
* normal renal function (serum creatinine ≤ 200 μmol/l)

Exclusion Criteria:

* pregnancy
* lack of written concent
* emergency operation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 410 (Actual)
Dates: Start 2010-12; Primary Completion 2012-07 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Clinical outcome quantified by using the Sequential Organ Failure Assessment (SOFA) Score | 3 days

SECONDARY OUTCOMES:
length of ICU stay in hours | outcome at 28 days
incidence of acute renal failure | 28 days
total requirement of vasoconstrictors | 28 days
total requirement of fluid replacement therapy | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Haberthuer, MD, Principal Investigator — Anästhesie/chirurgische Intensivstation Luzerner Kantonsspital
Locations (3):
- Switzerland (3):
  - Kantonsspital Luzern, Lucerne, Canton of Lucerne
  - Departement of Anaesthesia and Intensive Care, University Hospital of Basel, Basel
  - Kantonsspital Luzern, Lucerne

REFERENCES:
- [Derived] Schmidt T, Pargger H, Seeberger E, Eckhart F, von Felten S, Haberthur C. Effect of high-dose sodium selenite in cardiac surgery patients: A randomized controlled bi-center trial. Clin Nutr. 2018 Aug;37(4):1172-1180. doi: 10.1016/j.clnu.2017.04.019. Epub 2017 May 2. PMID 28502744